CLINICAL TRIAL: NCT07263529
Title: Risk of Anemia Development and Clinical Effects of Oral Iron Therapy in Women (18-55 Years) With Non-Anemic Iron Deficiency
Brief Title: Risk of Anemia and Effects of Oral Iron Therapy in Non-Anemic Iron-Deficient Women (18-55 Years)
Acronym: NAID-F
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Osman Demir, MD, MD, Istanbul University - Cerrahpasa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-KAEK-22; E-14028348-302.14.02-985103 (Other: Istanbul Univ. Cerrahpasa Fac. of Medicine); E-15916306-604.01-281470566 (Other: Istanbul Provincial Health Directorate)
Record Dates: First submitted 2025-11-16; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Non-Anemic Iron Deficiency
Keywords: Iron deficiency without anemia; Risk of anemia; Clinical effects of oral iron therapy; Women 18-55; Ferritin; Hemoglobin; Symptom scores; Nutritional intervention; Iron supplementation
MeSH Terms: conditions — Iron Deficiencies | interventions — Diet Therapy; ferrous sulfate

STUDY DESIGN:
Intervention Model Description: All participants initially receive the same nutritional intervention; after post-intervention evaluation, subgroups are defined and those with persistent iron deficiency receive the drug intervention.
Masking Description: No parties are masked; this is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARM 1 - Nutritional Intervention with Post-Intervention Subgrouping (Experimental): All participants (N=60) begin with isolated non-anemic iron deficiency and receive a 2-month standardized nutritional intervention to improve iron intake and absorption. Afterward, participants are stratified into five subgroups (ARM1-0 to ARM1-4) based on hematologic response. Subgroups ARM1-1 to ARM1-4 represent persistent deficiency (ferritin <15 µg/L with normal CRP) and will receive oral elemental iron.
  * ARM1-0: Normalized or maintained iron status (no deficiency) - no iron therapy administered.
  * ARM1-1: Persistent isolated iron deficiency - receives oral elemental iron.
  * ARM1-2: Minimal hemoglobin decline (<1 g/dL) with microcytosis/hypochromia - receives oral elemental iron.
  * ARM1-3: Hemoglobin decline >1 g/dL but above anemia threshold, with microcytosis/hypochromia - receives oral elemental iron.
  * ARM1-4: Overt iron deficiency anemia - receives oral elemental iron.
  Interventions: Other: Dietary Intervention (2 months); Drug: Oral Elemental Iron (Ferrous Sulfate) 80 mg/day

INTERVENTIONS:
Other: Dietary Intervention (2 months) — A two-month nutritional counseling program for all participants (N = 60) with isolated non-anemic iron deficiency. The program emphasized the inclusion of iron-rich foods (both heme and non-heme sources), the use of enhancers of iron absorption (such as vitamin C), and practical strategies to reduce absorption inhibitors (e.g., limiting tea and coffee consumption around meals, reviewing antacid use). Participants received biweekly phone follow-ups to monitor adherence and assess symptoms.
  Other Names: Nutritional Intervention (2 months)
Drug: Oral Elemental Iron (Ferrous Sulfate) 80 mg/day — One-month oral therapy with 80 mg elemental iron (ferrous sulfate) daily for participants with persistent iron deficiency after the nutritional phase (ferritin < 15 µg/L). Biweekly phone follow-up for adherence and symptom checks. Adherence and side effects monitored at clinic visit or by phone.
  Other Names: Oral Iron Intervention (1 month)

SUMMARY:
This study investigates the risk of anemia development in women aged 18-55 years with non-anemic iron deficiency and evaluates the clinical effects of oral iron therapy. The study consists of a two-month nutritional intervention phase followed by a one-month oral iron treatment phase. Participants first receive dietary counseling aimed at increasing iron intake and absorption. After two months, changes in hematologic parameters and symptoms are evaluated. Women with persistent iron deficiency then receive daily oral ferrous sulfate (80 mg elemental iron) for one month. The study aims to identify early predictors of anemia progression and to assess the impact of dietary modification and oral iron therapy on symptoms and laboratory findings.

DETAILED DESCRIPTION:
This study examines the risk of anemia development in women aged 18-55 years with non-anemic iron deficiency (NAID) and evaluates the clinical effects of oral iron therapy in those with persistent deficiency. The objective is to characterize individual and clinical factors associated with progression toward anemia and to assess the impact of nutritional modification and subsequent iron supplementation on hematologic and symptom-based outcomes.

Iron deficiency is one of the most common nutritional deficiencies globally. NAID often remains unrecognized despite its potential to cause fatigue, decreased physical performance, and progression to anemia if untreated. Iron plays a key role in oxygen transport, DNA synthesis, and muscle metabolism. Dietary intake includes both heme (animal-derived) and non-heme (plant-derived) forms with differing bioavailability. Ferritin is the primary biomarker used to diagnose iron deficiency, though inflammatory conditions may influence its accuracy. A careful differential evaluation is important to distinguish NAID from other causes of anemia such as chronic disease, B12 or folate deficiency, thalassemia syndromes, thyroid disorders, or gastrointestinal blood loss.

The study uses a two-phase, single-center prospective design at Kağıthane 5 No'lu Family Health Center (ASM), Istanbul, Turkey, conducted under ethics committee approval and institutional permission. In the initial two-month observational phase, participants receive standardized dietary counseling aimed at increasing iron intake and improving absorption. Health status and adherence are monitored biweekly. After this period, participants are categorized into four groups according to hematologic changes: isolated iron deficiency; microcytosis/hypochromia with minimal hemoglobin decline (<1 g/dL) ; greater hemoglobin decline without meeting anemia thresholds; or overt iron deficiency anemia.

In the subsequent one-month experimental phase, participants with persistent deficiency receive oral ferrous sulfate providing 80 mg elemental iron daily. Clinical and laboratory evaluations are performed at designated time points to assess changes in complete blood count parameters, ferritin, serum iron indices, inflammatory markers, and patient-reported symptoms.

Primary outcomes include changes in symptom scores, while secondary outcomes evaluate hematologic and biochemical responses. Planned analyses explore associations between baseline characteristics, dietary habits, and anemia progression. Power analysis using repeated measures ANOVA indicated a required sample size of 60 participants.

This research highlights the importance of individualized management strategies for iron deficiency, aiming to support appropriate use of supplementation while reducing unnecessary treatment and potential adverse effects. Enhancing dietary iron intake may help prevent anemia progression, promote patient safety, and improve resource utilization in primary care settings.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 18-55 years (including premenopausal and menopausal women).
* Normal hemoglobin level (≥ 12 g/dL).
* Serum ferritin < 15 μg/L (WHO criteria for iron deficiency).
* Mentzer index > 13.
* Normal levels of vitamin B12, folic acid, thyroid hormones (TSH and sT4), and C-reactive protein (CRP < 5 mg/L).
* Non-anemic iron deficiency confirmed by laboratory results.
* Good general health and cognitive capacity to provide informed consent.
* Willingness to participate, comply with study procedures, and provide written informed consent.

Exclusion Criteria:

* Pregnancy or postpartum period.
* Acute or chronic infections.
* History or suspicion of malignancy.
* Chronic inflammatory or autoimmune diseases.
* Chronic fatigue syndrome or depressive disorders.
* Chronic kidney disease or renal failure (acute or chronic).
* Congestive heart failure, ischemic heart disease, or cerebrovascular disease.
* Coagulopathy or clinically significant bleeding tendency.
* Hematological disorders (e.g., thalassemia, hemoglobinopathies).
* Postoperative patients, transplant recipients, or dialysis patients.
* Currently using any form of iron supplementation or treatment.
* Any condition that, in the investigator's opinion, may interfere with the participant's safety or the interpretation of study results.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Patient-Reported Iron Deficiency Symptom Scores After 2-Month Nutritional Intervention and 1-Month Oral Iron Therapy | Baseline, Week 8 (post-nutritional intervention), Week 12 (post-oral iron therapy)
  Change in patient-reported symptoms including fatigue, weakness, dizziness, and cognitive function etc. measured at baseline, after 2-month nutritional intervention, and after 1-month oral iron therapy.

SECONDARY OUTCOMES:
Change from Baseline in Hemoglobin and Red Blood Cell Indices After 2-Month Nutritional Intervention and 1-Month Oral Iron Therapy | Baseline, Week 8, Week 12
  Hemoglobin, hematocrit, MCV, MCH, MCHC, and ferritin measured at baseline, Week 8, and Week 12.
Change from Baseline in Serum Iron and Total Iron Binding Capacity After 2-Month Nutritional Intervention and 1-Month Oral Iron Therapy | Baseline, Week 8, Week 12
  Serum iron, TIBC, and ferritin measured at baseline, Week 8, and Week 12.
Incidence of Progression to Anemia After 2-Month Nutritional Intervention | Baseline to Week 8
  Number and proportion of participants who progress from non-anemic iron deficiency (baseline Hb ≥12 g/dL) to anemia (Hb <12 g/dL) measured at Week 8 (post-nutritional intervention). This outcome assesses the short-term risk of anemia development despite dietary counseling focused on iron-rich foods and absorption enhancement.
Proportion of Participants Demonstrating Hematologic Response to 1-Month Oral Iron Therapy (Hb increase ≥1.0 g/dL) | Week 8 to Week 12
  Proportion of participants with an increase in hemoglobin ≥1.0 g/dL between Week 8 (pre-treatment) and Week 12 (post-treatment). Hematologic response defined as hemoglobin increase ≥1.0 g/dL after 1-month oral ferrous sulfate (80 mg/day elemental iron) therapy.
Proportion of Participants Demonstrating Ferritin Response to 1-Month Oral Iron Therapy (Ferritin increase ≥15 µg/L or ≥30 µg/L absolute) | Week 8 to Week 12
  Proportion of participants with ferritin increase ≥15 µg/L from Week 8 to Week 12, or achieving ferritin ≥30 µg/L at Week 12. Biochemical response reflecting iron store replenishment after oral iron therapy, measured by increase in serum ferritin.

OTHER OUTCOMES:
Adherence to Nutritional Intervention Over 2 Months | Week 0 to Week 8
  Participant adherence to dietary counseling measured via food logs and biweekly phone calls.
Adherence to Oral Iron Therapy Over 1 Month | Week 8 to Week 12
  Compliance with daily oral iron (ferrous sulfate 80 mg/day) assessed by pill count and self-report.
Incidence of Treatment-Related Adverse Events During 1-Month Oral Iron Therapy | Week 8 to Week 12
  Gastrointestinal or other adverse events reported during oral iron therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Osman Demir, MD, Principal Investigator — Kağıthane No.5 Family Health Center, Istanbul, Turkey; Ayşen Fenercioğlu, Assoc Prof, Study Director — Istanbul University - Cerrahpaşa, Cerrahpaşa Faculty of Medicine
Locations (1):
- Kagıthane No. 5 Family Health Center, Kâğıthane, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ortancil O, Sanli A, Eryuksel R, Basaran A, Ankarali H. Association between serum ferritin level and fibromyalgia syndrome. Eur J Clin Nutr. 2010 Mar;64(3):308-12. doi: 10.1038/ejcn.2009.149. Epub 2010 Jan 20. PMID 20087382
- [Background] Skolmowska D, Glabska D, Kolota A, Guzek D. Effectiveness of Dietary Interventions to Treat Iron-Deficiency Anemia in Women: A Systematic Review of Randomized Controlled Trials. Nutrients. 2022 Jun 30;14(13):2724. doi: 10.3390/nu14132724. PMID 35807904
- [Result] Silva Neto LGR, Santos Neto JED, Bueno NB, de Oliveira SL, Ataide TDR. Effects of iron supplementation versus dietary iron on the nutritional iron status: Systematic review with meta-analysis of randomized controlled trials. Crit Rev Food Sci Nutr. 2019;59(16):2553-2561. doi: 10.1080/10408398.2018.1459469. Epub 2018 Apr 30. PMID 29611716
- [Result] Moretti D, Goede JS, Zeder C, Jiskra M, Chatzinakou V, Tjalsma H, Melse-Boonstra A, Brittenham G, Swinkels DW, Zimmermann MB. Oral iron supplements increase hepcidin and decrease iron absorption from daily or twice-daily doses in iron-depleted young women. Blood. 2015 Oct 22;126(17):1981-9. doi: 10.1182/blood-2015-05-642223. Epub 2015 Aug 19. PMID 26289639
- [Result] Stefan MW, Gundermann DM, Sharp MH, Jennings BA, Gheith RH, Lowery RP, LowDog T, Ghatak SB, Barbosa J, Wilson JM. Assessment of the Efficacy of a Low-Dose Iron Supplement in Restoring Iron Levels to Normal Range among Healthy Premenopausal Women with Iron Deficiency without Anemia. Nutrients. 2023 Jun 3;15(11):2620. doi: 10.3390/nu15112620. PMID 37299583
- [Result] Nemeth E, Ganz T. Hepcidin and Iron in Health and Disease. Annu Rev Med. 2023 Jan 27;74:261-277. doi: 10.1146/annurev-med-043021-032816. Epub 2022 Jul 29. PMID 35905974
- [Result] Zhu XY, Wu TT, Wang HM, Li X, Ni LY, Chen TJ, Qiu MY, Shen J, Liu T, Ondo WG, Wu YC. Correlates of Nonanemic Iron Deficiency in Restless Legs Syndrome. Front Neurol. 2020 Apr 30;11:298. doi: 10.3389/fneur.2020.00298. eCollection 2020. PMID 32425874
- [Result] Sawada T, Konomi A, Yokoi K. Iron deficiency without anemia is associated with anger and fatigue in young Japanese women. Biol Trace Elem Res. 2014 Jun;159(1-3):22-31. doi: 10.1007/s12011-014-9963-1. Epub 2014 Apr 23. PMID 24756645
- [Result] da Silva Lopes K, Yamaji N, Rahman MO, Suto M, Takemoto Y, Garcia-Casal MN, Ota E. Nutrition-specific interventions for preventing and controlling anaemia throughout the life cycle: an overview of systematic reviews. Cochrane Database Syst Rev. 2021 Sep 26;9(9):CD013092. doi: 10.1002/14651858.CD013092.pub2. PMID 34564844
- [Result] Miles LF, Litton E, Imberger G, Story D. Intravenous iron therapy for non-anaemic, iron-deficient adults. Cochrane Database Syst Rev. 2019 Dec 20;12(12):CD013084. doi: 10.1002/14651858.CD013084.pub2. PMID 31860749
- [Result] Houston BL, Hurrie D, Graham J, Perija B, Rimmer E, Rabbani R, Bernstein CN, Turgeon AF, Fergusson DA, Houston DS, Abou-Setta AM, Zarychanski R. Efficacy of iron supplementation on fatigue and physical capacity in non-anaemic iron-deficient adults: a systematic review of randomised controlled trials. BMJ Open. 2018 Apr 5;8(4):e019240. doi: 10.1136/bmjopen-2017-019240. PMID 29626044
- [Result] Fletcher A, Forbes A, Svenson N, Wayne Thomas D; A British Society for Haematology Good Practice Paper. Guideline for the laboratory diagnosis of iron deficiency in adults (excluding pregnancy) and children. Br J Haematol. 2022 Feb;196(3):523-529. doi: 10.1111/bjh.17900. Epub 2021 Oct 24. No abstract available. PMID 34693519
- [Result] Clenin GE. The treatment of iron deficiency without anaemia (in otherwise healthy persons). Swiss Med Wkly. 2017 Jun 14;147:w14434. doi: 10.4414/smw.2017.14434. eCollection 2017. PMID 28634965
- [Result] WHO guideline on use of ferritin concentrations to assess iron status in individuals and populations [Internet]. Geneva: World Health Organization; 2020. Available from http://www.ncbi.nlm.nih.gov/books/NBK569880/ PMID 33909381
- [Result] Balendran S, Forsyth C. Non-anaemic iron deficiency. Aust Prescr. 2021 Dec;44(6):193-196. doi: 10.18773/austprescr.2021.052. Epub 2021 Dec 1. PMID 35002031
- [Result] Guideline on haemoglobin cutoffs to define anaemia in individuals and populations [Internet]. Geneva: World Health Organization; 2024. Available from http://www.ncbi.nlm.nih.gov/books/NBK602198/ PMID 38530913
- [Result] Soppi ET. Iron deficiency without anemia - a clinical challenge. Clin Case Rep. 2018 Apr 17;6(6):1082-1086. doi: 10.1002/ccr3.1529. eCollection 2018 Jun. PMID 29881569
- See also: Ethical approval: Istanbul University-Cerrahpasa Clinical Research Ethics Committee. — https://etikkurul.iuc.edu.tr/tr/iletisim
- See also: Study site: Kagithane 5 No'lu Family Health Center (ASM), conducted by Dr. Osman Demir. — https://www.kagithane5noluasm.com.tr/
- See also: Institutional authorization: Permission for study implementation obtained from Istanbul Provincial Health Directorate. — https://istanbulism.saglik.gov.tr/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-10-28): https://cdn.clinicaltrials.gov/large-docs/29/NCT07263529/Prot_SAP_000.pdf
  • Informed Consent Form (2025-10-28): https://cdn.clinicaltrials.gov/large-docs/29/NCT07263529/ICF_001.pdf